CLINICAL TRIAL: NCT04461379
Title: Prevention, Efficacy and Safety of BCG Vaccine in COVID-19- Randomized Clinical Trial
Brief Title: Prevention, Efficacy and Safety of BCG Vaccine in COVID-19 Among Healthcare Workers
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, René Rodríguez-Gutiérrez, Professor Endocrinology Division, Facultad de Medicina, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EN20-00011
Record Dates: First submitted 2020-07-02; First posted 2020-07-08 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: BCG; COVID-19; SARS-CoV2; Corona Virus Infection
Keywords: Healthcare workers
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — BCG Vaccine

STUDY DESIGN:
Intervention Model Description: A randomized double-blinded clinical trial, using computer software, participants will be allocated between two groups:
  Intervention: BCG vaccine intradermally 0.1 ml, equivalent to 0.075 mg of attenuated Mycobacterium bovis. (Tokio 172 strain). The application technique is based on the National Vaccination Manual version 2017.
  Comparator: Placebo, intradermally 0.1 ml of NaCl 0.9%
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, researchers (including members of the research team that will assess outcomes), and treating physicians or health personnel (should the patient require in-hospital management) will be blinded to the treatment group to which the patients were randomized. Only the personnel who apply the vaccine will not be blinded to the treatment group to which the patients were randomized (this personnel will not have any further contact with the patients or provide any other type of patient care).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCG Vaccine (Experimental): A single dose BCG vaccine intradermally 0.1 ml.
  Interventions: Biological: BCG vaccine
- Placebo (Placebo Comparator): A single dose intradermally 0.1 ml of NaCl 0.9% solution
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: BCG vaccine — A single dose BCG vaccine intradermally (deltoid region of the right arm) 0.1 ml, equivalent to 0.075 mg of attenuated Mycobacterium bovis . (Tokio 172 strain)
  Other Names: Calmette-Guerin Bacillus vaccine
  Arms: BCG Vaccine
Other: Placebo — A single dose intradermally ((deltoid region of the right arm) 0.1 ml of NaCl 0.9% solution
  Arms: Placebo

SUMMARY:
In Mexico the total number of confirmed cases of COVID-19 is 232, 000 and 28,510 deaths. Health workers are at high risk of COVID-19 infection. Their absence from work dramatically limits the ability to contain the disease. There is currently no vaccine to prevent the disease. Since the introduction to the vaccination schedule of the Bacillus Calmette-Guerin (BCG) live attenuated vaccine directed towards tuberculosis prevention, a decrease in infant mortality has been reported, not related only to tuberculosis. BCG vaccine has been hypothesized to have a non-specific role towards other unrelated pathogens such as viruses that cause airway disease, with reduced morbidity and mortality. In murine as well as in human models it has been shown to decrease the incidence of acute respiratory influenza infections. Likewise, in countries with a high endemicity for tuberculosis, the BCG vaccine reduces the incidence of respiratory infections by up to 80% . In healthy subjects, the BCG vaccine increases the production of proinflammatory cytokines in monocytes. Likewise, it increases the epigenetic response, causing an increase in the transcription of genes important in the antimicrobial response, as well as an improvement in cellular function. This is the first national clinical trial to evaluate prospectively the effect that the BCG vaccine offers towards the prevention and reduction of severity in cases of COVID-19.

DETAILED DESCRIPTION:
The study design is a randomized, double-blinded, placebo-controlled clinical trial.

Age stratified randomization (<45 years and> 45 years) was performed using permuted blocks with allocation concealment.

The sample size is 908 patients. 454 patients in each stratum (227 with placebo and 227 with BCG vaccine).

Eligible participants will be healthcare professionals over 18 years of age who are in contact with patients with COVID-19, with negative IgG and IgM antibodies results for SARS-CoV-2 prior to their inclusion and sign the informed consent. After signing the informed consent, the participants will be randomized 1:1 to the intervention group (BCG vaccine) or control (placebo), a medical history will be performed, and a blood plasma sample will be obtained to determine specific antibodies against SARS-CoV-2.

The patients will be followed up for 6 months after the application of the vaccine, they will be contacted by phone every two weeks in order to identify the adverse effects of the vaccine (30 days after the application) as well as to identify symptoms of COVID-19, in addition, follow-up visits will be carried out at the third and sixth months, in each of these visits a blood plasma sample will be obtained and IgG and IgM antibodies will be measured.

Statistical Analysis Type: By intention to treatment

ELIGIBILITY:
Inclusion Criteria:

* Health workers who are working onsite in patients' areas with COVID-19
* Age > 18 years
* Negative specific IgG and IgM antibodies test result for SARS CoV-2 before the enrollment.
* Provide a signed and dated informed consent form

Exclusion Criteria:

* Age <18 years
* Positive test for specific antibodies IgG and IgM antibodies result for SARS Cov-2
* Primary or secondary immunosuppression
* Use of immunosuppression drugs, use of hydroxychloroquine, cloroquine, Azithromycin, Lopinavir/ritonavir, Ivermectin or any other drug used to treat patients COVID-19 before the enrollment.
* Chemotherapy treatment
* Presence of antibodies IgA, IgM, IgG against SARS-CoV-2
* Pregnancy or breastfeeding
* Missing informed consent form
* Fever > 38° in the previous 24 hours
* Any BCG vaccine contraindication
* History of previous allergy to the components of the vaccine
* Already part of any other trial
* Previous or active tuberculosis (TB) disease
* Another vaccine administrated 4 months before the start of the trial.
* Any underlying history of malignancy or lymphoma.
* Actual treatment with steroids
* Absence of more than 1 month from the hospital, from the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 908 (Estimated)
Dates: Start 2020-07-21 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Demonstrate COVID- 19 disease incidence among Health care workers: | During the 6 months study period
  Cumulative incidence of infection in 6 months:
  disease defined as positive SARS-Cov-2 test (serology), plus fever (using self-reported questionnaire), or at least one sign or symptom of respiratory disease including cough, shortness of breath, respiratory distress/failure (using self-reported questionnaire)
Demonstrate cumulative incidence of hospitalization for COVID-19 among Health care workers: | During the 6 months study period
  Cumulative incidence of hospitalization for COVID-19
Demonstrate the Incidence of specific Antibodies against SARS-CoV-2 at 3 and 6 months in health care workers | During the 6 months study period
  Incidence of specific Antibodies (IgG and IgM) against SARS-CoV-2 will be measured at 3 and 6 months
Hospitalization of severe disease COVID-19 | During the 6 months study period
  Number of participants who needed hospitalization
Oxygen supplementation in severe disease COVID-19 | During the 6 months study period
  Number of participants who Need for oxygen supplementation (nasal cannulas, masks, high flow oxygen) in hospitalized patients
Need for intubation or non-invasive ventilation for the patient. | During the 6 months study period
  Number of participants who Need for intubation or non-invasive ventilation in hospitalized patients
Critical care admission with SARS-CoV2 | During the 6 months study period
  Number of participants in Critical care admission with SARS-CoV2 in hospitalized patients
Mortality associated to progressive pulmonary disease | During the 6 months study period
  Mortality associated to progressive pulmonary disease in hospitalized patients

SECONDARY OUTCOMES:
Evaluate the safety of the vaccine by measuring the incidence rates of local and systemic adverse effects that occur after one month its application. | 1 month after vaccine/placebo application
Calculate the incidence of COVID-19 complications | During the 6 months study period
Determine the mean days of hospitalization and days in intensive care unit by COIVD-19 | During the 6 months study period
Calculate the cost associated with in-hospital medical care | During the 6 months study period
Determine the scores of the Clinical Prediction Rules associated with mortality using Sequential Organ Failure Assessment (SOFA score) at the patient's hospital admission: | During the 6 months study period
  SOFA score: PaO2/FIO2 (mm Hg), SaO2/FIO2, Platelets (×10³/µL), Bilirubin (mg/dL), Hypotension, Glasgow Coma Score and Creatinine (mg/dL) or urine output (mL/d).
Determine the scores of the Clinical Prediction Rules associated with mortality using Acute Physiology and Chronic Health disease Classification System (APACHE) at the patient's hospital admission: | During the 6 months study period
  APACHE: History of severe organ failure or immunocompromise Heart Failure Class IV, cirrhosis, chronic lung disease, or dialysis-dependent, Age, Temperature (C°), Mean arterial pressure (mmHg), pH, Sodium (mEq/L), Potassium (mEq/L), Creatinine (mg/dL), Hematocrit (%), WBC (x 109/L)
Evaluate and determine the alteration profile in laboratory studies at the patient's hospital admission | During the 6 months study period
  CPR, ESR, Ferritin, D-dimer, LDH,Troponins, Procalcitonin, Interleukin-6, Hemoglobin, Hematocrit, Erythrocytes, Leukocytes, MCV, HCM, MCHC, Lymphocytes, Monocytes, Eosinophils, Basophils, Platelets, Glucose, Urea, Creatinine, BUN, Sodium, Potassium, Chlorine, Calcium, Serum albumin, Direct bilirubin, Indirect bilirubin, Alkaline phosphatase, AST, ALT, bleeding time, Prothrombin Time, Activated partial thromboplastin time, Arterial / Venous Blood Gasometry, pH, pCO2, HCO3, pO2, SaO2%, Lactate.
Registration of chronic medications | During the 6 months study period
Need for vasopressors | During the 6 months study period

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario "José E. González", Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.who.int/emergencies/diseases/novel-coronavirus-2019
- See also: Related Info — http://www.nature.com/articles/s41585-020-0325-9
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/32393823
- See also: Related Info — https://www.gob.mx/salud%7Ccensia/documentos/manual-de-vacunacion-edicion-2017